CLINICAL TRIAL: NCT01732393
Title: Effect of Quercetin in Prevention and Treatment of Chemotherapy Induced Oral Mucositis in Blood Dyscrasias
Brief Title: Effect of Quercetin in Prevention and Treatment of Oral Mucositis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Pegah Mosannen Mozafari, assistant professor of oral medicine, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 89470
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Chemotherapy Induced Oral Mucositis
Keywords: Quercetin; Chemotherapy; Mucositis; Hematologic Malignancies
MeSH Terms: conditions — Mucositis; Hematologic Neoplasms | interventions — Quercetin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oral quercetin capsules (Active Comparator): Patients in the intervention group were administered two, 250 mg Quercetin capsules daily for 3 weeks
  Interventions: Drug: oral quercetin capsules
- oral placebo capsules (Placebo Comparator): Patients in the placebo group received two placebo capsules containing lactose .
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: oral quercetin capsules — 10 cases in case group and 10 cases in control group. Patients in the intervention group were administered two, 250 mg Quercetin capsules daily for 3 weeks. Patients in the placebo group received two placebo capsules containing lactose .Patients were examined every other day for evaluation of initiation and severity of oral mucositis.
  Arms: oral quercetin capsules
Drug: Placebo
  Arms: oral placebo capsules

SUMMARY:
The study aims to evaluate the effect of Quercetin (a natural flavonoid) on prevention of and treatment of chemotherapy-induced oral mucositis in patients with blood malignancies.

ELIGIBILITY:
Inclusion Criteria:

* patient under chemotherapy
* for a hematologic malignancy
* the hematologist permits the trial on the patient
* agreement of patient for participating in the trial

Exclusion Criteria:

* presence pf ANY oral lesion at the beginning of the trial
* loss of follow up
* use of digoxin and cyclosporine
* patient death

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
lower grade of mucositis | 3 weeks
  grade of mucositis due to WHO criteria

SECONDARY OUTCOMES:
duration of mucositis | 3 weeks of study tiem span and after trial
  duration of mucositis due to Who criteria

CONTACTS AND LOCATIONS:
Overall Officials: Pegah Mosannen Mozafari, assistant professor, Study Director — Mashhad University of Medical Sciences
Locations (1):
- Oral Medicine Department of Mashhad dental School, Mashhad, Khorasan Razavi, Iran